CLINICAL TRIAL: NCT06364475
Title: Comparing the Effects of Time-restricted Eating and Three Meals-three Snacks Diet on Body Composition and on Biochemical Parameters
Brief Title: Could a Time-restricted Diet Compete With a Calorie-restricted 6-meal Diet?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Aclan Özder, Professor, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BezmialemVU-TF-AÖ-1
Record Dates: First submitted 2024-04-04; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Nutrition Therapy; Weight Loss; Intermittent Fasting
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: One group 16:8 time-restricted intermittent fasting and the other group energy-restricted six-meal eating. Both of groups with an eating plan suitable with their groups and 400 kcal lower than the total daily energy requirement and with similar macronutrient content (50% carbohydrates, 25% fat and 25% protein).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16:8 Time-Restricted Intermittent Fasting Group (Active Comparator): 88 people were included in the 16:8 time-restricted intermittent fasting group with an 8-hour window for food consumption, with an eating plan of 400 kcal lower than the total daily energy requirement.
  Interventions: Behavioral: 16:8 Time-Restricted Intermittent Fasting Group
- Energy-Restricted Six-Meal Group (Active Comparator): 86 people were included in the energy-restricted six-meal group. This group have an eating plan three meal and three snack of 400 kcal lower than the total daily energy requirement.
  Interventions: Behavioral: Energy-Restricted Six-Meal Group

INTERVENTIONS:
Behavioral: 16:8 Time-Restricted Intermittent Fasting Group — Participants total daily energy expenditures were calculated using the Harris-Benedict formula. This group have a feeding window 8 hours and eating plan of 400 kcal lower than the total daily energy requirement and with similar macronutrient content (50% carbohydrates, 25% fat and 25% protein). Participants in the time-restricted eating group were allowed to drink calorie-free. They were expected to follow their diet for two months during the study.
  Arms: 16:8 Time-Restricted Intermittent Fasting Group
Behavioral: Energy-Restricted Six-Meal Group — Participants total daily energy expenditures were calculated using the Harris-Benedict formula. This group have an eating plan three meals and three snacks of 400 kcal lower than the total daily energy requirement and with similar macronutrient content (50% carbohydrates, 25% fat and 25% protein). They were expected to follow their diet for two months during the study.
  Arms: Energy-Restricted Six-Meal Group

SUMMARY:
The prevalence of obesity and obesity-related diseases are on the rise worldwide. The widely accepted approach in dietary treatment of obesity is the calorie-restricted three meals-three snacks a day diet; however, alternative approaches are needed. This study was conceived with a view to comparing time-restricted eating, a method which can be easily conveyed and applied in overcoming obesity, to a six meals a day diet. 174 participants aged between 18-65 with a BMI>25 kg/m2 were included. Diet lists with similar calorie, macro counts suitable for their respective group were prepared. Anthropometric measurements, blood pressure, blood tests were analyzed before the study and at the end of the 8-week.

DETAILED DESCRIPTION:
Our study was conducted with participants, aged between 18-65 and with a BMI >25 kg/m2, who consulted a family medicine clinic in Istanbul, accepted the terms and conditions of the study and signed the volunteer consent form. Sample analysis was performed by T.M. with G Power 3.1.9.7 (Franz Faul, Germany), using data from Sundfør et al.'s study, "Effect of intermittent versus continuous energy restriction on weight loss, maintenance and cardiometabolic risk: a randomized 1-year trial". The effect size was assumed to be d: 0.382 for the purposes of calculation. After the calculation made with the aforementioned effect size, with 80% power and 10% margin of error, it was concluded that a cohort of at least 126 samples, of which 63 would be in the patient group and 63 would be in the control group, should be used in this study.

People with a history of bariatric surgery, eating disorders, alcohol and drug addiction, anti-obesity medication use, diagnosed with diabetes and hypothyroidism, active cancer patients and people carrying infectious diseases were excluded from the study. At the beginning of the study, 88 people were included in the 16:8 time-restricted intermittent fasting (time-restricted eating) group, with an eating plan of 400 kcal lower than the total daily energy requirement and with similar macronutrient content (50% carbohydrates, 25% fat and 25% protein); and 86 people were included in the energy-restricted six-meal group. Diet lists suitable for each group were prepared, and food substitution lists were handed out to the participants. Control measurements were performed after the 4th week. In order to keep the participants' motivation high throughout the study, an online chat group with the participation of a physician and dietitian, was set up. The study was concluded with 137 patients, because 37 people had left the study by the end of 8 weeks. Total daily energy expenditures were calculated using the Harris-Benedict formula. Participants in the time-restricted eating group were allowed to drink calorie-free soda, unsweetened tea, herbal tea and coffee during their 16-hour fast.

Anthropometric measurements, blood pressure measurements, as well as fasting blood glucose, ALT (alanine aminotransferase), AST (aspartate aminotransferase), lipid panel and HbA1c values in blood samples were checked at the start and the end of the study. Body composition was measured with the bioelectric impedance method with a Tanita Compacto CS 601. The bioelectrical impedance method is prone to error because of fluctuations in body water content. However, it is accepted as a valid method for assessing changes in weight loss studies when duly accompanied by X-ray absorptiometry and reference methods suitable for evaluating multi-compartment body composition under standard conditions [14]. Waist circumference, waist-to-hip ratio and waist-to-height ratio (WHtR), which is recently being recommended, correlate better than BMI in assessing the obesity-related health burden , including total mortality rate, type 2 diabetes, and CVD (cardiovascular disease) risk. The CBC (complete blood count) tests were performed with a Mindrat BC-6800 device, using the SF Cube technology; biochemical tests were performed with a Roche Cobas C702 device that works with photometry; and HbA1c tests were performed with an Arkray HA-8180V device that performs measurements based on the HPLC (High-Performance Liquid Chromatography) technique.

All statistical analyses were performed with the help of SPSS (Statistical Package for the Social Sciences) v. 25.0. The conformity of variables to the normal distribution pattern were checked with histogram graphics and Kolmogorov-Smirnov test. Average, standard deviation, median, IQR (Inter Quantile Range), min.-max. values were used while presenting defining analyses. Categorical variables were compared with Pearson Chi Square Test. Mann Whitney U Test was used in examining the nonparametric variants between groups. The Wilcoxon Test was used for assessing the change in the monitored values within a group, and Repeated Measures Analysis was used for the same purpose when the comparison was being made between the groups. Cases where the P value was under 0.05 were taken as statistically significant results.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65
* BMI >25 kg/m2

Exclusion Criteria:

* People with a history of bariatric surgery
* Eating disorders
* Alcohol and drug addiction
* Anti-obesity medication use
* Diagnosed with diabetes and hypothyroidism
* Active cancer patients
* People carrying infectious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Weight measured in kilogram | Two months
  It contains weight measured in kilogram. This was measured with Tanita Compacto CS 601 which one 0.1 kg sensitive scale.

SECONDARY OUTCOMES:
Body composition | Two months
  Body composition was measured with the bioelectric impedance method with a Tanita Compacto CS 601. The bioelectrical impedance method is prone to error because of fluctuations in body water content. However, it is accepted as a valid method for assessing changes in weight loss studies when duly accompanied by X-ray absorptiometry and reference methods suitable for evaluating multi-compartment body composition under standard conditions.
Body mass index | Two months
  The BMI is calculated by dividing an adult's weight in kilograms by their height in metres squared. It is expressed in units of kg/m2.
Waist-to-height ratio (WHtR) | Two months
  The waist-height ratio is calculated as waist measurement divided by height measurement, in centimeters.
Waist circumference in centimetres | Two months
  Waist value was measured at the apex of the iliac crest as recommended by the United States National Institutes of Health.

CONTACTS AND LOCATIONS:
Overall Officials: Aclan Ozder, Prof, Study Director — Bezmialem Vakif University
Locations (1):
- İstanbul Sabri Artam Vakfi Family Medicine Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If they need my data, they can contact me by e-mail.